CLINICAL TRIAL: NCT03734926
Title: A Phase 1, Open-Label, Dose-Escalation and Expansion, Safety and Tolerability Study of ZSP1241 in Participants With Advanced Solid Tumors
Brief Title: A Phase 1 Study of ZSP1241 in Participants With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Zhongsheng Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZSP1241-18-01
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinoma; Cholangiocarcinoma; Gastric Cancer; Esophageal Cancer; Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Stomach Neoplasms; Esophageal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Participants with advanced solid tumors including hepatocellular carcinoma, cholangiocarcinoma, gastric cancer, esophageal cancer, colorectal cancer and other advanced solid tumors.
  Interventions: Drug: ZSP1241
- Part 2 Cohort A (Experimental): Participants with hepatocellular carcinoma.
  Interventions: Drug: ZSP1241
- Part 2 Cohort B (Experimental): Participants with gastric cancer, esophageal cancer, colorectal cancer and other advanced solid tumor.
  Interventions: Drug: ZSP1241

INTERVENTIONS:
Drug: ZSP1241 — ZSP1241 tablets for oral administration.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics, and determine the maximum tolerated dose of ZSP1241 in participants with hepatocellular carcinoma, cholangiocarcinoma, gastric cancer, esophageal cancer, colorectal cancer and other advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants are required to meet all the criteria below in order to be included in the trial:

  1. Male or female patient, aged 18 ~ 75 years.
  2. Confirmed diagnosis of advanced solid tumors by histological or cytological examination, participants have no effective standard anticancer therapy available or is intolerant to standard anticancer therapy.
  3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
  4. Participants with at least 1 measurable tumor lesion based on RECIST 1.1.
  5. Recovery from past medical history of adverse reactions (excluding alopecia and neurotoxicity) caused by radiotherapy and/or chemotherapy to NCI CTCAE 5.0 Grade ≤ 1 or baseline level.
  6. Life expectancy ≥ 12 weeks.
  7. Adequate organ function, defined by the following laboratory results, to be obtained prior to enrollment:

     Bone marrow function: ANC≥1.5×109/L; HB≥90 g/L; PLT≥75×109/L. Liver function: ALT≤2.5×ULN, AST≤2.5×ULN, ALP≤2.5×ULN, TBIL≤1.5×ULN; ALT≤5×ULN, AST≤5×ULN (For participants with liver focal masses and metastasis).

     Renal function: creatinine≤1.5×ULN; CL≥ 50 mL/min. Coagulation function: INR≤1.5×ULN; INR≤2.3×ULN (For participants with liver focal masses and metastasis).
  8. Child-Pugh class A (only for hepatocellular carcinoma and cholangiocarcinoma).
  9. Participants (including partners) who have no gestation plans and are willing to follow reliable contraceptive measures during the study and until 8 months after the last dosing.
  10. Participants with voluntarily signature Informed Consent Form (ICF) prior to screening.

Exclusion Criteria:

* Eligible participants must not meet any of the following exclusion criteria:

  1. Participants who have intracranial tumor and/or brain metastases with clinical symptoms needed treatment are ineligible not including the following :

     1. recovery from the therapy (including radiotherapy and/or surgery) 4 weeks before enrollment.
     2. participants with intracranial tumor who are clinically stable during screening and enrollment, no need to medication by hormone or anticonvulsants, and predicted to be clinically stable during the study.
  2. Participants who suffer from chronic and active infective diseases and require systemic antibiotic, antifungal, or antiviral treatment except concomitant antiviral systemic therapy for chronic hepatitis B or C.
  3. Participants with dysphagia.
  4. Participants with incontrollable hydrops in third lumen such as malignant pleural effusion and ascites.
  5. Participants with history of pulmonary fibrosis or interstitial pneumonia including pneumoconiosis and radiation pulmonary fibrosis beyond radiation field.
  6. Participants who suffer from irritable bowel syndrome and need medication.
  7. Participants with any clinically significant gastrointestinal abnormalities such as Crohn's disease, ulcerative colitis and subtotal gastrectomy.
  8. Participants with major surgery in recent 4 weeks or active peptic ulcer disease or unrecovered wound.
  9. Participants with history of myocardial infarction or congestive heart-failure (CHF) at NYHA≥3 level within 6 months prior to enrollment.
  10. Participants with LVEF<50% during screening.
  11. Participants with QTcF prolongations in ECG baseline ( QTcF>450ms for males or QTcF>470ms for females) or high risk factors leading to QT intervals prolonging (including hypokalemia, familial QT interval prolongation syndrome) or a history of uncontrollable blood pressure or a history of severe or uncontrollable ventricular arrhythmia such as two or three degree atrioventricular block.
  12. Participants with medications known as QTc prolongation or TDP ventricular tachycardia inducer or strong inhibitors and inducers of CYP3A4 not less than 5 days or 5 half-times before first dosing ZSP1241.
  13. Participants with history of most recently chemotherapy, radiotherapy, or non-antibody antitumor biologics within 4 weeks prior to the first ZSP1241 treatment and last time medication of nitrosoureas, mitomycin C or doxorubicin within 6 weeks and latest usage of antibody antitumor biologics within 4 weeks.
  14. Participants with current or prior retinal detachment or presently confirmed diagnosis keratopathy including but not limited to bullous keratopathy, calcific band keratopathy, corneal abrasion, keratohelcosis, keratitis and so on.
  15. Participants with history of autoimmune disease.
  16. Pregnant or nursing women.
  17. Participants who, in the judgment of the investigator, will be unfit for the study. ( For reasons such as poor compliance, unsuitable for venous catheterization and so on)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of ZSP1241 in single dose ascending (SAD) and multiple dose ascending (MAD) as measured by assessment of maximum tolerated dose (MTD), dose limiting toxicity (DLT) and treatment emergent adverse events (TEAEs) | At Day 7 for SAD Part and At day 28 after for MAD part
  Participant with TEAEs assessed by CTCAE V5.0

SECONDARY OUTCOMES:
Time to progression (TTP). | Screening, Day 28 of Cycle 1 (28 days), then every 6 weeks for hepatocellular carcinoma or 8 weeks for other advanced solid tumors, until disease progression or discontinuation from study (up to 18 months).
Overall response rate (ORR). | Screening, Day 28 of Cycle 1 (28 days), then every 6 weeks for hepatocellular carcinoma or 8 weeks for other advanced solid tumors, until disease progression or discontinuation from study (up to 18 months).
Cmax of ZSP1241 | Protocol-defined time points during Cycles 0 (7 days) and 1 (28 days) of treatment per subject.
  Defined as maximum observed plasma concentration
Tmax of ZSP1241 | Protocol-defined time points during Cycles 0 (7 days) and 1 (28 days) of treatment per subject.
  Defined as time to maximum plasma concentration
Cmin of ZSP1241 | Protocol-defined time points during Cycles 0 (7 days) and 1 (28 days) of treatment per subject.
  Defined as minimum observed plasma concentration during the dosing interval
AUC0-t of ZSP1241 | Protocol-defined time points during Cycles 0 (7 days) and 1 (28 days) of treatment per subject.
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration
t½ of ZSP1241 | Protocol-defined time points during Cycles 0 (7 days) and 1 (28 days) of treatment per subject.
  Defined as the apparent plasma terminal phase disposition half-life
Cl/F of ZSP1241 | Protocol-defined time points during Cycles 0 (7 days) and 1 (28 days) of treatment per subject.
  Defined as oral dose clearance

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China